CLINICAL TRIAL: NCT06436950
Title: Electrical Phrenic Nerve Stimulation in Patients With Ventilator-induced Diaphragm Dysfunction: a Randomized Controlled Study
Brief Title: Electrical Phrenic Nerve Stimulation in Patients With VIDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Wang Zongyu, Principal Investigator, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEPNS_01
Record Dates: First submitted 2024-05-20; First posted 2024-05-31 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-06

CONDITIONS: Diaphragms; Phrenic Nerves
Keywords: Ventilator-induced diaphragmatic dysfunction; transcutaneous electrical phrenic nerve stimulation

STUDY DESIGN:
Intervention Model Description: Transcutaneous electrical phrenic nerve stimulation (TEPNS) group: TEPNS+usual care Control group: usual care
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- transcutaneous electrical phrenic nerve stimulation (TEPNS) group (Experimental): The patients in TEPNS group receive TEPNS and usual care.
  Interventions: Device: transcutaneous electrical phrenic nerve stimulation (TEPNS)
- Control group (No Intervention): The patients in control group receive usual care only.

INTERVENTIONS:
Device: transcutaneous electrical phrenic nerve stimulation (TEPNS) — TEPNS is conducted twice a day for consecutive 5 days. Electrodes are applied to bilateral neck skin which phrenic nerve runs underneath.
  Arms: transcutaneous electrical phrenic nerve stimulation (TEPNS) group

SUMMARY:
This study aims to examine efficacy of transcutaneous electrical phrenic nerve stimulation (TEPNS) in ventilator-induced diaphragmatic dysfunction (VIDD). The investigators recruit VIDD patients, and randomly assign the patients into TEPNS group and control group. TEPNS group receives TEPNS twice a day for consecutive 5 days. Control group only receives usual care. The investigators collect diaphragm function indicators and outcomes to evaluate the efficacy.

DETAILED DESCRIPTION:
Ventilator-induced diaphragmatic dysfunction (VIDD) is common in intensive care unit (ICU). There is a need of measurements to improve VIDD. The investigators hypothesize that transcutaneous electrical phrenic nerve stimulation (TEPNS) will increase diaphragmatic function. This study is a single centre, randomized controlled trial with control or treatment group in a 1:1 ratio. Eligible patients include aged ≥ 18 years, ventilated for at least 48 h with an expected stay of more than 7 days in the ICU, and diaphragm thickening fraction (DTF)< 25%. The patients are randomly allocated to either receiveTEPNS and usual care (TEPNS group) or usual care only (control group). Blind is not used. TEPNS is conducted twice a day for consecutive 5 days. Electrodes are applied to bilateral neck skin which phrenic nerve runs underneath. Clinical data are collected, including baseline characteristics, airway pressure, esophageal pressure, gastric pressure, ventilation days, ICU length of stay, 28-day mortality, etc.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years
* ventilated for at least 48 h with an expected stay of more than 7 days in the ICU
* diaphragm thickening fraction (DTF)< 25%

Exclusion Criteria:

* having a pacemaker
* cutaneous lesion that could interfere with probes
* previous diaphragmatic nerve paralysis
* body mass index > 35 kg/m2
* severe chronic obstructive pulmonary disease (FEV1/FVC<30%)
* pregnancy or lactation
* decision to withhold life-sustaining treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Transdiaphragmatic pressure (Pdi) | Collected once a day after transcutaneous electrical phrenic nerve stimulation (TEPNS) for consecutive 5 days
  Pdi=gastric pressure - esophageal pressure

SECONDARY OUTCOMES:
Airway pressure, esophageal pressure, gastric pressure, airway occlusion pressure, driving pressure, transpulmonary pressure | Collected once a day after TEPNS for consecutive 5 days
  Determined from respiratory mechanics indicators provided by ventilator or calculated from them
Esophageal pressure-time product | Collected once a day after TEPNS for consecutive 5 days
  Determined from respiratory mechanics indicators provided by ventilator
Ventilation days | Collected at 28 days after enrollment
  Mechanical ventilation days in 28 days after enrollment
Length of ICU stay | Collected at 28 days after enrollment
  Days of ICU stay in 28 days after enrollment
28-day mortality | Collected at 28 days after enrollment
  Survival outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Zongyu Wang, Dr., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Bao Q, Chen L, Chen X, Li T, Xie C, Zou Z, Huang C, Zhi Y, He Z. The effects of external diaphragmatic pacing on diaphragm function and weaning outcomes of critically ill patients with mechanical ventilation: a prospective randomized study. Ann Transl Med. 2022 Oct;10(20):1100. doi: 10.21037/atm-22-4145. PMID 36388825
- [Background] Medrinal C, Machefert M, Lamia B, Bonnevie T, Gravier FE, Hilfiker R, Prieur G, Combret Y. Transcutaneous electrical diaphragmatic stimulation in mechanically ventilated patients: a randomised study. Crit Care. 2023 Aug 30;27(1):338. doi: 10.1186/s13054-023-04597-1. PMID 37649092
- [Background] O'Rourke J, Sotak M, Curley GF, Doolan A, Henlin T, Mullins G, Tyll T, Omlie W, Ranieri MV. Initial Assessment of the Percutaneous Electrical Phrenic Nerve Stimulation System in Patients on Mechanical Ventilation. Crit Care Med. 2020 May;48(5):e362-e370. doi: 10.1097/CCM.0000000000004256. PMID 32191413
- [Background] Sotak M, Roubik K, Henlin T, Tyll T. Phrenic nerve stimulation prevents diaphragm atrophy in patients with respiratory failure on mechanical ventilation. BMC Pulm Med. 2021 Oct 8;21(1):314. doi: 10.1186/s12890-021-01677-2. PMID 34625059
- [Background] Poulard T, Bachasson D, Fosse Q, Nierat MC, Hogrel JY, Demoule A, Gennisson JL, Dres M. Poor Correlation between Diaphragm Thickening Fraction and Transdiaphragmatic Pressure in Mechanically Ventilated Patients and Healthy Subjects. Anesthesiology. 2022 Jan 1;136(1):162-175. doi: 10.1097/ALN.0000000000004042. PMID 34788380
- [Background] Goligher EC, Dres M, Patel BK, Sahetya SK, Beitler JR, Telias I, Yoshida T, Vaporidi K, Grieco DL, Schepens T, Grasselli G, Spadaro S, Dianti J, Amato M, Bellani G, Demoule A, Fan E, Ferguson ND, Georgopoulos D, Guerin C, Khemani RG, Laghi F, Mercat A, Mojoli F, Ottenheijm CAC, Jaber S, Heunks L, Mancebo J, Mauri T, Pesenti A, Brochard L. Lung- and Diaphragm-Protective Ventilation. Am J Respir Crit Care Med. 2020 Oct 1;202(7):950-961. doi: 10.1164/rccm.202003-0655CP. PMID 32516052